CLINICAL TRIAL: NCT03655821
Title: Individualized Pemetrexed Dosing in Patients With Non-small Cell Lung Cancer or Mesothelioma Based on Renal Function to Improve Treatment Response
Brief Title: Dose Individualization of Pemetrexed - IMPROVE-II
Acronym: IMPROVE-II
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 81 patients included, difficult inclusion and full inclusion would not change the results
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPROVE-II
Record Dates: First submitted 2018-05-14; First posted 2018-08-31 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Non Small Cell Lung Cancer; Mesothelioma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (BSA-based dosing) (Active Comparator): Dosing of pemetrexed is based on BSA according drug label
  Interventions: Drug: Pemetrexed
- Arm B (renal function based dosing) (Experimental): Dosing of pemetrexed is based on renal function, calculated to reach the target AUC.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Dosing is either based on BSA or renal function

SUMMARY:
Rationale:

Pemetrexed is a multi-targeted folate antagonist, which is primarily indicated for the treatment of advanced non-small cell lung cancer (NSCLC) and mesothelioma. Dosing of cytotoxic agents like pemetrexed requires balancing the dual risk of sub-therapy and toxicity. Administration of pemetrexed to patients with a creatinine clearance <45 ml/min is currently not advised. Pemetrexed is dosed based on body surface area (BSA), while renal function and dose are the sole determinants for systemic exposure. This causes 3 major issues:

1. In patients with renal dysfunction, BSA-based dosing may lead to haematological toxicity
2. Patients have to discontinue treatment due to declining renal function, and are withheld effective treatment
3. Even in patients with adequate renal function (GFR >45 ml/min) treatment may be improved by individualized dosing based on renal function, resulting in less toxicity. Also, BSA-based dosing may lead to ineffective therapy in patients with above average renal function.

The investigators aim to address these problems.

Objective: The overall main objective is to develop a safe and effective individualized dosing regimen for pemetrexed.

Study design: IMPROVE-II is an open label, double arm, randomized study to compare renal function-based dosing of pemetrexed versus BSA-based dosing on attainment of therapeutic exposure.

Study population: IMPROVE-II includes 94 patients with NSCLC or mesothelioma that are eligible for pemetrexed treatment.

Intervention: patients will be randomized in a 1:1 ratio to Arm A (BSA-based dosing according drug label) or to Arm B (renal function based dosing). The renal function-based dose will be calculated to reach the target AUC. Pharmacokinetic assessment after administration will be performed after the first pemetrexed dose in both arms.

Main study endpoints: The fraction (percentage) of patients with attainment of therapeutic exposure with BSA-based dosing versus renal function-based dosing.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The investigators consider the extra burden from participating in the planned studies limited. The extra interventions compared to routine care, consist of sampling extra blood. The pharmacokinetic assessments require placement of one additional intravenous catheter. To ensure minimal impact of study participation on daily life, a limited sampling strategy will be used. Patients may benefit from participating in IMPROVE I and -II, as they will be treated with a potentially safe and effective drug that is dosed individually, which prevents toxic exposure.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Eligible for treatment with pemetrexed-based chemotherapy
3. Creatinine clearance >45ml/min
4. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
5. Subject is able and willing to sign the Informed Consent Form

Exclusion Criteria:

1. Conditions that affect haemostasis in a way that blood drawing is complicated (to be assessed by physician)
2. Contraindications for treatment with pemetrexed in line with the summary of product characteristics (SmPC) (except for creatinine clearance <45 ml/min in IMPROVE-I)

   1. Hypersensitivity to the active substance or to any of the excipients
   2. Pregnancy or lactation
   3. Concomitant yellow fever vaccine
3. The presence of clinically relevant pharmacokinetic interactions, according to the current SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Exposure (AUC) | 24 hours
  mg*h/l
The fraction (percentage) of patients with attainment of therapeutic exposure with BSA-based dosing versus renal function-based dosing. | 3 months
  The fraction (percentage) of patients with attainment of therapeutic exposure defined as an AUC of 164 mg*h/l ±25%, with pemetrexed dosing based on renal function versus BSA-based dosing.

SECONDARY OUTCOMES:
Population Clearance (Cl) | 3 months
  L/h
Population Intercompartmental Clearance (Q) | 3 months
  L/h
Population Central Volume of Distribution (V1) | 24 hours
  L
Population Peripheral Volume of Distribution (V2) | 3 months
  L
Performance of different renal function algorithms to predict pemetrexed | 3 months
  Significant change in objective function value (OFV) (<3.84 with 1 degree of freedom)
Performance of different renal function algorithms to predict pemetrexed pharmacokinetics (decrease in variability) | 3 months
  Decrease in clearance variablity (%)
Hematologic assessment during dosing based on renal function in patients with a creatinine clearance >45ml/min versus dosing based on BSA. | 5 days
  Complete blood count (no per liter)
The incidence of hematologic dose limiting toxicities (DLT) and adverse events, as measured with the CTCAE V4' | 3 months
  through listing
The incidence of non-hematologic dose limiting toxicities (DLT) and adverse events, as measured with the CTCAE V4 | 3 months
  through listing
The incidence of toxicity-related dose reductions, treatment delays and treatment discontinuation | 3 months
  through listing
Quality of life measured with the EORTC QLQ-C30/L13 questionnaire | 3 months
  0-100 scale
In silico evaluation of neutropenic response | 1 year
  Simulation of risk for neutropenic response
Neutropenia related costs | 1 year
  Euros

CONTACTS AND LOCATIONS:
Overall Officials: Rob ter Heine, PhD, Principal Investigator — Radboud University Medical Center
Locations (5):
- Netherlands (5):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Antoni van Leeuwenhoek, Amsterdam
  - Maastricht University Medical centre, Maastricht
  - Radboud university medical centre, Nijmegen
  - Erasmus University Medical Centre, Rotterdam

REFERENCES:
- [Derived] de Rouw N, Boosman RJ, Burgers JA, Huitema ADR, Dingemans AC, Derijks HJ, Burger DM, Piet B, Hendriks LEL, Biesma B, Pruis MA, Dumoulin DW, Croes S, Mathijssen RHJ, van den Heuvel MM, Ter Heine R. Renal function-based versus standard dosing of pemetrexed: a randomized controlled trial. Cancer Chemother Pharmacol. 2023 Jan;91(1):33-42. doi: 10.1007/s00280-022-04489-1. Epub 2022 Nov 21. PMID 36413252
- [Derived] Boosman RJ, de Rouw N, Huitema ADR, Burgers JA, Ter Heine R. Prediction of the pharmacokinetics of pemetrexed with a low test dose: A proof-of-concept study. Br J Clin Pharmacol. 2023 Feb;89(2):699-704. doi: 10.1111/bcp.15520. Epub 2022 Sep 21. PMID 36053283
- [Derived] de Rouw N, de Boer M, Boosman RJ, van den Heuvel MM, Burger DM, Lieverse JE, Derijks HJ, Frederix GWJ, Ter Heine R. The Pharmacoeconomic Benefits of Pemetrexed Dose Individualization in Patients With Lung Cancer. Clin Pharmacol Ther. 2022 May;111(5):1103-1110. doi: 10.1002/cpt.2529. Epub 2022 Feb 21. PMID 35048355